CLINICAL TRIAL: NCT06970431
Title: Effects of Preoperative Education Combined With Intraoperative Music Therapy on Perioperative Anxiety and Pain in Elective Cesarean Section Patients
Brief Title: Therapy on Perioperative Anxiety and Pain in Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCHH_012
Record Dates: First submitted 2025-04-08; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Music Therapy; Anxiety; Health Education
MeSH Terms: conditions — Anxiety Disorders; Health Education

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- reoperative Education + Intraoperative Music Therapy Arm (Experimental): The standardized preoperative education and the individualized music therapy during the operation are implemented jointly, and the patients' perioperative anxiety values, pain scores, shivering index, etc. are collected.
  Interventions: Other: eoperative Education + Intraoperative Music Therapy Arm
- Preoperative Education Alone Arm (Active Comparator): The control group only received standardized preoperative education.
  Interventions: Other: Preoperative Education Alone Arm

INTERVENTIONS:
Other: eoperative Education + Intraoperative Music Therapy Arm — The experimental group implemented standardized preoperative education one day before the operation (covering knowledge such as the surgical procedure), headphone fitting one hour before the operation (with a volume of 45-55 decibels), and music therapy throughout the operation and for 30 minutes after the operation (parturients can choose personalized music). Full-time nurses were responsible for the preoperative education, and trained operating room nurses implemented the music therapy. Meanwhile, data such as anxiety scores, pain scores, shivering index, postoperative complications, postoperative recovery status, and satisfaction surveys were collected at multiple time points through standardized tools.
  Arms: reoperative Education + Intraoperative Music Therapy Arm
Other: Preoperative Education Alone Arm — The control group received the same standardized preoperative education by full-time nurses one day before the operation, covering surgical procedures, precautions, anesthesia, and postoperative recovery.
  Data were collected at multiple time points using standardized tools, including anxiety scores (before and 6, 12, 24 h after surgery via GAD-7), pain scores (before and 6, 12, 24 h after via VAS), shivering index (before surgery, before wearing headphones, when leaving OR), postoperative complications (wound infection, urinary retention, etc.), postoperative recovery indicators (time to get out of bed, anal exhaust, breastfeeding start, hospital stay), and satisfaction surveys (24 h after surgery).
  Importantly, the control group had no music therapy intervention before, during, or after surgery.
  Arms: Preoperative Education Alone Arm

SUMMARY:
This study aims to explore the effects of preoperative education combined with intraoperative music therapy on perioperative anxiety and pain in patients undergoing elective cesarean section. The study subjects were patients scheduled for cesarean section under combined spinal - epidural anesthesia. A prospective study design with random grouping was adopted. Through systematic preoperative education and intraoperative music intervention, multi - dimensional evaluations were carried out to analyze the effects of preoperative education combined with intraoperative music therapy on the relief of perioperative anxiety, pain and shivering in patients, as well as its impact on postoperative recovery and nursing satisfaction.

DETAILED DESCRIPTION:
I. Research Methods A prospective randomized controlled trial design will be used. Eligible elective cesarean patients will be randomly assigned to an experimental group (preoperative education + intraoperative music therapy) or a control group (routine preoperative education only).

1. Preoperative Health Education Conducted by dedicated nurses 1 day before surgery, covering surgical procedures, precautions, anesthesia, and postoperative recovery.
2. Intraoperative Music Therapy Experimental group: Headphones fitted 1 hour preoperatively at 45-55 decibels, playing personalized or pre-screened music continuously during surgery and for 30 minutes postoperatively.

   Intervention timing: Headphone adaptation and volume adjustment 1 hour preoperatively; continuous playback during surgery; 30-minute playback postoperatively to reduce anxiety and discomfort.

   Executors: Preoperative education by specialized nurses; music therapy by trained operating room nurses to ensure equipment and volume stability.
3. Data Collection

   Assessments at specified time points using standardized tools:

   Anxiety: GAD-7 scale (preoperative, 6h, 12h, 24h postoperatively). Pain: VAS scale (preoperative, 6h, 12h, 24h postoperatively). Shivering index: Cold Shivering Index Scale (preoperative, before headphone use, at discharge from the operating room).

   Postoperative complications: Wound infection, urinary retention, hemorrhage, heart failure, or pulmonary embolism.

   Recovery indicators: Ambulation time, anal exhaust time, lactation time, hospital stay.

   Satisfaction surveys: Nursing and anesthesia satisfaction via questionnaires 24h postoperatively.
4. Study Population

Inclusion criteria:

18-40 years old, singleton pregnancy, eligible for elective cesarean section. No severe pregnancy complications (e.g., preeclampsia, gestational diabetes). Able to provide informed consent and complete follow-ups.

Exclusion criteria:

Complications or diseases affecting study outcomes. Severe mental illness preventing protocol understanding. Refusal to participate or incomplete follow-ups. Allergy to music/headphones. II. Technical Route Literature review & protocol design: Develop the study plan and obtain ethical approval.

Patient recruitment & randomization: Enroll patients per criteria; use random number tables for grouping.

Intervention & data recording: Standardized interventions by the research team; regular data verification.

Data analysis & reporting: Statistical analysis to compare group differences; summarize findings and draft reports.

III. Feasibility Analysis Sample size: Estimated 64 patients per group (140 total, including 10% dropout rate) based on anxiety score differences and literature.

Ethical feasibility: Informed consent obtained; complies with ethical review requirements.

Technical feasibility: Hospital equipped with nursing tools (headphones, assessment scales) and a skilled team.

Resource feasibility: Reasonable budget and 10-month timeline ensure timely data collection, analysis, and reporting.

ELIGIBILITY:
Inclusion Criteria： ASA grade I or II, aged 18-40 years female must be singleton pregnancy eligible

Exclusion Criteria:

History of pregnancy-related complications severe pregnancy complications (e.g., preeclampsia, gestational diabetes mellitus) Severe mental illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
anxiety score | Baseline, up to 12 hours postoperatively, up to 24 hours postoperatively
  Before the operation and at 6 hours, 12 hours, and 24 hours after the operation, the Generalized Anxiety Disorder 7-item scale (GAD-7 scale) is used.The Generalized Anxiety Disorder 7-Item Scale (GAD-7) is a widely used tool to assess the severity of generalized anxiety symptoms.
  Score Range: Scores range from 0 to 21, with each of the 7 items rated on a 4-point scale (0 = "Not at all" to 3 = "Nearly every day").
  Interpretation: Higher scores indicate worse outcomes, reflecting more severe anxiety symptoms. Specifically:
  0-4: Minimal anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety This scale helps clinicians and researchers quantify anxiety levels, with higher scores signifying greater distress and functional impairment.
pain score | Baseline, up to 12 hours postoperatively, up to 24 hours postoperatively
  The Visual Analogue Scale (VAS) is used to assess pain intensity. Full Name: Visual Analogue Scale Score Range: Scores range from 0 to 10, where 0 = "No pain" and 10 = "Worst pain imaginable".
  Interpretation: Higher scores indicate worse outcomes, reflecting more severe pain.
  Assessment Time Points: Pain is evaluated at preoperative baseline, and at 6 hours, 12 hours, and 24 hours postoperatively to measure acute pain changes during the perioperative period.
  This validated single-item scale allows patients to rate their pain on a continuous numeric scale, providing a straightforward method to quantify pain severity. Clear time-specific assessments (preoperative and postoperative time points) ensure standardized data collection for comparing intervention effects between groups.

SECONDARY OUTCOMES:
shivering index | baseline (before any intervention is initiated), Immediately After Birth,Perioperative
  The Cold Shivering Index Scale (CSIS) is used to evaluate the severity of intraoperative shivering. Scores range from 0 to 4, with specific criteria:
  0 = No shivering
  1. = Faint shivering (visible muscle contraction without body movement)
  2. = Mild shivering (mild, controlled body movement)
  3. = Moderate shivering (obvious body tremors affecting the surgical field)
  4. = Severe shivering (uncontrollable whole-body shaking interfering with surgery).
  Higher scores indicate worse outcomes, reflecting more severe shivering and decreased patient comfort during surgery.
Record of postoperative complications | Complications during hospitalization(assessed up to 5 days)
  Such as wound infection, urinary retention, bleeding, heart failure or pulmonary embolism, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Study Director — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Na Li , MD, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No